CLINICAL TRIAL: NCT00163501
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 3 Clinical Trial to Assess the Long Term Safety of Ciclesonide, Applied as a Nasal Spray (200 Mcg, Once Daily) in the Treatment of Perennial Allergic Rhinitis (PAR) in Patients 12 Years and Older
Brief Title: Safety and Effectiveness of Ciclesonide Nasal Spray in Patients With Perennial Allergic Rhinitis During One Year Treatment (BY9010/M1-404)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-404
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Perennial Allergic Rhinitis; Allergic Rhinitis; Hay Fever
Keywords: Allergy; Perennial Allergic Rhinitis; Allergic Rhinitis; Hay Fever
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Hypersensitivity | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of ciclesonide nasal spray as compared with placebo (inactive substance) nasal spray in relieving symptoms of perennial allergic rhinitis.

ELIGIBILITY:
Main Inclusion Criteria:

* General good health, other than perennial allergic rhinitis
* History and diagnosis of perennial allergic rhinitis by skin prick test

Main Exclusion Criteria:

* Participation in any investigational drug trial within the 30 days preceding the Screening Visit
* A known hypersensitivity to any corticosteroid or any of the excipients in the formulation
* Use of any prohibited concomitant medications as defined by the study protocol

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2003-12; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
change in Total Nasal Symptom Scores.

SECONDARY OUTCOMES:
change in symptoms, quality of life, safety.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (39):
- United States (39):
  - Altana Pharma/Nycomed, Encinitas, California
  - Altana Pharma/Nycomed, Huntington Beach, California
  - Altana Pharma/Nycomed, Long Beach, California
  - Altana Pharma/Nycomed, Los Angeles, California
  - Altana Pharma/Nycomed, Mission Viejo, California
  - Altana Pharma/Nycomed, Newport Beach, California
  - Altana Pharma/Nycomed, San Diego, California
  - Altana Pharma/Nycomed, Stockton, California
  - Altana Pharma/Nycomed, Vista, California
  - Altana Pharma/Nycomed, Trumbull, Connecticut
  - Altana Pharma/Nycomed, Clearwater, Florida
  - Altana Pharma/Nycomed, DeLand, Florida
  - Altana Pharma/Nycomed, Atlanta, Georgia
  - Altana Pharma/Nycomed, Normal, Illinois
  - Altana Pharma/Nycomed, Overland Park, Kansas
  - Altana Pharma/Nycomed, New Orleans, Louisiana
  - Altana Pharma/Nycomed, Bethesda, Maryland
  - Altana Pharma/Nycomed, North Dartmouth, Massachusetts
  - Altana Pharma/Nycomed, Forked River, New Jersey
  - Altana Pharma/Nycomed, Skillman, New Jersey
  - Altana Pharma/Nycomed, Springfield, New Jersey
  - Altana Pharma/Nycomed, Liverpool, New York
  - Altana Pharma/Nycomed, Raleigh, North Carolina
  - Altana Pharma/Nycomed, Winston-Salem, North Carolina
  - Altana Pharma/Nycomed, Cincinnati, Ohio
  - Altana Pharma/Nycomed, Oklahoma City, Oklahoma
  - Altana Pharma/Nycomed, Portland, Oregon
  - Altana Pharma/Nycomed, Easton, Pennsylvania
  - Altana Pharma/Nycomed, Pittsburgh, Pennsylvania
  - Altana Pharma/Nycomed, Cranston, Rhode Island
  - Altana Pharma/Nycomed, Austin, Texas
  - Altana Pharma/Nycomed, Dallas, Texas
  - Altana Pharma/Nycomed, Houston, Texas
  - Altana Pharma/Nycomed, Kerrville, Texas
  - Altana Pharma/Nycomed, New Braunfels, Texas
  - Altana Pharma/Nycomed, San Antonio, Texas
  - Altana Pharma/Nycomed, Salt Lake City, Utah
  - Altana Pharma/Nycomed, Richmond, Virginia
  - Altana Pharma/Nycomed, Milwaukee, Wisconsin

REFERENCES:
- See also: BY9010-M1-404-RDS-2005-12-11.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4532&filename=BY9010-M1-404-RDS-2005-12-11.pdf